CLINICAL TRIAL: NCT03230149
Title: Prevalence and Characteristics of Fabry Disease (FD) in Patients With Stroke or Small Fiber Neuropathy
Acronym: FABRY
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Shire International GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: HAO16026
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Fabry Disease
Keywords: Fabry; Stroke; Cerebrovascular Accident; small fiber neuropathy
MeSH Terms: conditions — Fabry Disease; Stroke; Small Fiber Neuropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Molecular and genetic tests: Measurements of the alpha-GAL enzyme activity will be performed knowing that for male patients with alpha-GAL activities below the cut-off value and all female patients, a blood sampling for full genetic sequencing of all seven exons including promotors of the a-GAL gene will be done
  Interventions: Diagnostic Test: Measurements of the alpha-GAL enzyme activity

INTERVENTIONS:
Diagnostic Test: Measurements of the alpha-GAL enzyme activity — Blotting paper blood tests in order to highlight an enzyme deficiency for hemizygous males with DBS kits in order to detect Fabry disease, with genetic confirmation if an abnormality is detected. For women genotyping is mandatory.

SUMMARY:
FD is pan-ethnic. Its reported annual incidence of 1 in 100,000 may underestimate the true prevalence of the disease. Indeed, recently, in addition with affected males FD developing a "classic" phenotype, " cardiac variant " and " renal variant " have been reported for FD patients with predominant or exclusive cardiac or renal involvement. " Neurologic variant " could exist.

Nervous system can be affect by FD leading to cerebrovascular diseases (ischemic or haemorrhagic strokes, TIA (Transient Ischemic Attacks) or peripheral neuropathy (acroparesthesias and pain).

Aims will be to determine the prevalence of Fabry disease in patients with stroke or small fiber neuropathy, and their characteristics

DETAILED DESCRIPTION:
FD is pan-ethnic. Its reported annual incidence of 1 in 100,000 may underestimate the true prevalence of the disease. Indeed, recently, in addition with affected males FD developing a "classic" phenotype, " cardiac variant " and " renal variant " have been reported for FD patients with predominant or exclusive cardiac or renal involvement. " Neurologic variant " could exist.

Nervous system can be affect by FD leading to cerebrovascular diseases (ischemic or haemorrhagic strokes, TIA (Transient Ischemic Attacks) or peripheral neuropathy (acroparesthesias and pain).

1. Considering strokes, they are the third leading cause of death in France, with more than 140,000 people presenting a stroke per year. Stroke incidence is 1-2/1000 people per year. If the mean age of stroke patient is 72 yo, 25% of them are under 55 yo. The etiology of stroke in young patients remains undetermined in up to half of the cases. Data on prevalence of FD in people with cryptogenic ischaemic stroke are limited and controversial. In addition to cryptogenic strokes, FD can lead to stroke from arterial or heart diseases (secondary to high blood pressure, renal insufficiency, cardiomyopathy, rate variability, arrhythmias, valvular insufficiency).

   The investigators aimed to evaluate the frequency of FD in a cohort of stroke patients in tertiary stroke centers in consecutively recruited patients under 60 yo. The investigators will include patients with so-called cryptogenic stroke but also stroke patients due to large artery atherosclerosis, cardioembolism, and small-vessel occlusion. The investigators will also study the clinical and radiological characteristic of stroke patients due to FD, and will compare these data with those from patients without FD, supported by biochemical and genetic findings.
2. Considering peripheral nervous system, Small fiber neuropathy (SFN) is a subgroup of peripheral neuropathy which is characterized by an affection of the thin myelinated A-δ and unmyelinated C-fibers. SFN patients present with sensory symptoms and pain. SFN are not a rare condition; recent study showed a minimum prevalence of 50/100.000. The most commonly etiology reported for SFN is diabetes mellitus ; Other possible etiologies include connective tissue disease, celiac disease, thyroid dysfunction, vitamin B12 deficiency, monoclonal gammopathy, HIV and hepatitis C infections, amyloidosis, toxicity due to alcohol or drugs, and hereditary neuropathies including FD, suspected to be underdiagnosed.

In SFN patients,the investigators aimed to screen for FD in our tertiary national center for peripheral neuropathies, in addition to others diseases or affections, to evaluate the frequency of FD in a large cohort of SFN patients, and describe the clinical phenotype of SFN in FD patients compared to other ones.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 yo and under 60 yo
* diagnosed with a TIA / stroke (ischemic and haemorrhagic strokes) based on clinical evaluation and MRI
* diagnosed with small fibers neuropathy (SFN) with normal nerve conduction studies in conventional electrophysiology

Exclusion Criteria:

* patients over 60 yo

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients between 18 and 60 years old diagnosed with a TIA/ strocke or a SFN
Sampling Method: Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
frequency of FD in a cohort of stroke patients | at the end of the study (an average of 2 years)
  number of patients with fabry disease in the cohort of stroke patients (1000 patients)

SECONDARY OUTCOMES:
frequency of FD in a cohort of Small fiber neuropathy (SFN) patients | at the end of the study (an average of 2 years)
  number of patients with fabry disease in the cohort of small fiber neuropathy patients (100 patients)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bicêtre, UNSIV (neurovascular stroke unit), Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No